CLINICAL TRIAL: NCT05276830
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy, and Safety Study of BXCL501 For The Treatment of Agitation Associated With Dementia
Brief Title: An Efficacy, and Safety Study Of BXCL501 For The Treatment Of Agitation Associated With Dementia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for business reasons; not due to safety or efficacy concerns
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXCL501-203
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Agitation; Dementia
MeSH Terms: conditions — Psychomotor Agitation; Dementia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Study will randomize subjects 1:1:1 to receive BXCL501 40 μg, BXCL501 60 μg, or matching placebo film
Who Masked: Participant, Investigator
Masking Description: Double-Blind, Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 40 micrograms (Experimental): Sublingual film containing 40 micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- 60 micrograms (Experimental): Sublingual film containing 60 micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Placebo (Experimental): Sublingual Placebo film
  Interventions: Drug: Placebo film

INTERVENTIONS:
Drug: BXCL501 — Sublingual film containing 40 Micrograms BXCL501
  Other Names: Dexmedetomidine
  Arms: 40 micrograms
Drug: BXCL501 — Sublingual film containing 60 Micrograms BXCL501
  Other Names: Dexmedetomidine
  Arms: 60 micrograms
Drug: Placebo film — Matching Sublingual Placebo film
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled parallel group 3-arm study assessing efficacy, safety, and tolerability of two doses BXCL501 in male and female geriatric residents (65 years and older) with acute agitation associated with all forms of dementia (i.e., probably Alzheimer's Disease, vascular dementia; mixed; frontotemporal dementia) excluding Parkinson's-Related Dementia and Lewy Body Dementia.

DETAILED DESCRIPTION:
The study will enroll at least 75 subjects to receive a single film consisting of BXCL501 40 μg dose, BXCL501 60 μg dose, or matching placebo film. Subjects must reside in a residential care facility and must require at least moderate assistance with activities of daily living (e.g., bathing, dressing, and toileting). The subject must be able to self-administer the film to participate in the study.

The effects of BXCL 501 on acute agitation will be assessed by the following scales: PEC, PAS, ACES, and CGI-I.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with any form of dementia (i.e., probable Alzheimer's Disease; vascular dementia; mixed; frontotemporal dementia)
2. Subjects who have met DSM-5 criteria for dementia (major neurocognitive disorder) who have instances of acute psychomotor agitation.
3. History of psychomotor agitation (e.g., kick, bite, flailing) to the point that it impairs social activities, requires staffing, or medical intervention, or impairs ability for functional activities of daily living.
4. Subjects are expected to exhibit behaviors that are congruent with the International Psychogeriatric Association criterion for agitation representing a change from the subject's usual behavior.
5. Subjects who have a score of ≤16 on the Mini-Mental State Exam (MMSE).
6. Subjects with a remote (>5 years) history of stroke may be included, regardless of size/location.
7. Subjects who read, understand, and provide written informed consent, or who have a legally authorized representative (LAR).
8. Subjects who are deemed to be medically appropriate for study participation by the principal investigator.
9. Subjects who are at their current location for at least 14 days before screening and plan to remain at the same location for the duration of the study.
10. Subjects who have the capability to participate in the study and self-administer the investigational product.
11. Subjects who are on a stable concomitant medications regimen for the treatment of any concurrent conditions for at least one month prior to the screening visit.

Exclusion Criteria:

1. Subjects who have dementia associated with Parkinson's disease and/or Lewy Body Disease are excluded.
2. Subjects suffering from alcohol and/or substance abuse.
3. Subjects with agitation caused by acute intoxication must be excluded.
4. Subjects with significant risk of suicide or homicide per the investigator's assessment.
5. Subjects who have hydrocephalus, seizure disorder, or history of significant head trauma, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, or focal neurological findings, with a recent (1 year) large (non-microvascular) stroke who may be considered medically unstable or in recovery must be excluded.
6. History of clinically significant syncope or syncopal attacks, orthostatic hypotension within the past 2 years.
7. Subjects with laboratory or ECG abnormalities.
8. Subjects with serious, unstable, or uncontrolled medical illnesses must be excluded.
9. Subjects who have received an investigational drug within 30 days prior to Screening must be excluded.
10. Subjects who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving dexmedetomidine must be excluded.
11. Subjects whose agitation is attributed to pain or infection, delirium, concomitant medications, environmental conditions, or another psychiatric condition or medical condition as determined by the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (3):
- United States (3):
  - Bioxcel Clinical Research Site, North Miami, Florida
  - Bioxcel Clinical Research Site, Springfield, Massachusetts
  - BioXcel Clinical Research Site, Toms River, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States from 08 February 2022 to 01 April 2022.
Groups:
- BXCL501: 40 Micrograms: Participants received a single sublingual film containing 40 micrograms Dexmedetomidine (BXCL501)
- BXCL501: 60 Micrograms: Participants received a single sublingual film containing 60 micrograms Dexmedetomidine (BXCL501)
- Placebo: Participants received a single sublingual matching placebo film
Period: Overall Study
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
Started | 2 | 1 | 2
Completed | 2 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 1 | 0 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 1 | 0 | 3
  Black or African American | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score
Description: The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: 120 minutes
Population: The study was terminated for business reasons, No data were collected for the outcome measures.
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline for Pittsburgh Agitation Scale
Description: The Pittsburgh Agitation Scale (PAS) assesses agitation for individuals with dementia across four behavior groups: aberrant vocalizations, motor agitation, aggressiveness, and resisting care. Each behavior group is scored ranging from 0 (not present) to 4 (maximally present).
Time Frame: 120 minutes
Population: The study was terminated for business reasons, No data were collected for the outcome measures.
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline for Agitation-Calmness Evaluation Scale
Description: The Agitation-Calmness Evaluation Scale (ACES) is a single item measure rating overall agitation and sedation, where 1 indicates marked agitation; 2 - moderate agitation; 3 - mild agitation; 4 - normal behavior; 5 - mild calmness; 6 - moderate calmness; 7 - marked calmness; 8 - deep sleep; and 9 - unarousable
Time Frame: 120 minutes
Population: The study was terminated for business reasons, No data were collected for the outcome measures.
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Clinical Global Impression - Improvement
Description: The Clinical Global Impression - Improvement (CGI-I) for agitation in response to treatment measures the current level of agitation relative to the level of agitation prior to administration of study intervention. The CGI-I scores range from 1 to 7 with a score of 1 indicating very much improved, and a score of 7 indicating very much worse.
Time Frame: 120 minutes
Population: The study was terminated for business reasons, No data were collected for the outcome measures.
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 7
Arm/Group | BXCL501: 40 Micrograms | BXCL501: 60 Micrograms | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BXCL501: 40 Micrograms (N=2) | BXCL501: 60 Micrograms (N=1) | Placebo (N=2)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to business reasons. There were no Safety or Efficacy Concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT05276830/Prot_SAP_000.pdf